CLINICAL TRIAL: NCT03881306
Title: CalliSpheres Drug-Eluting Beads With Oxaliplatin to Treat Inoperable NET Liver Metastases: A Multi-center Clinical Trial
Brief Title: DEBOXA for Inoperable NET Liver Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NET11330
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Neuroendocrine Tumors; Neoplasm Metastasis; Liver
Keywords: TACE; Oxaliplatin
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-TACE (Experimental): D-TACE for inoperable NEN liver metastases. Embolization agent: CalliSpheres Drug-Eluting Beads Chemotherapy agent: Oxaliplatin
  Interventions: Drug: D-TACE

INTERVENTIONS:
Drug: D-TACE — D-TACE with CalliSpheres-Oxaliplatin
  Other Names: CalliSpheres-Oxaliplatin

SUMMARY:
A prospective clinical trial to study the safety and effectiveness of Transcatheter Artery Chemotherapy and Embolization (TACE) using CalliSpheres Drug-Eluting Beads with oxaliplatin (DEBOXA) in treating patients who have inoperable neuroendocrine neoplasm (NEN) liver metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and effectiveness of Transcatheter Artery Chemotherapy and Embolization (TACE) using CalliSpheres Drug-Eluting Beads with oxaliplatin (DEBOXA) in patients with inoperable neuroendocrine neoplasm (NEN) liver metastases.

II. Determine the response rate (RR) of intrahepatic lesions in patients treated with this regimen.

III. Determine the overall survival (OS), progression-free survival time (DFS), time to hepatic progression (THP), and quality of life (QOL) in patients treated with this regimen.

IV. Safety assessment: adverse events (AEs) and severe adverse events(SAEs)

OUTLINE: This is a single-arm, multi-center, prospective study.

Patients receive D-TACE. Embolization agent: CalliSpheres Drug-Eluting Beads. Chemotherapy agent: oxaliplatin. Treatment repeats every 5 weeks in the absence of progression of hepatic lesions, or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis is confirmed by biopsy or clinical data, primary site is resected or primary site is not resected but without risks of bleeding, obstruction in the near future.
* Failure of ≥ 1 system treatment, such as long-acting somatostatin or EP chemotherapy regimen.
* Standard surgical resection can not be performed because of extent liver involvement （liver involvement ≥ 2 lobes or ≥ 2 major vessels）, or patients who are not willing to accept surgical operation.
* Predicted survival >3 months.
* Child Pugh Score: ≤ 7
* ECOG score for performance status: 0-1
* Informed consensus is achieved.

Exclusion Criteria:

* Metastases to other organs or sites besides liver.
* Prior TACE for liver tumors in 1 year.
* Obvious hepatic arterio-venous shunt or arterio-portal shunt.
* Prior or concurrent malignancy (Except basal carcinoma or squamous carcinoma of skin or carcinoma in situ of cervex uteri which has been cured).
* Platelet count < 50,000/mm^3 or white blood cell count <3,000 /mm^3 without hypersplenism.
* Creatinine greater than upper limit of normal (ULN)
* AST or AST > 5 times ULN
* Compromised coagulation: INR (International normalised ratio) >1.5, current anti-coagulation therapy or hemorrhagic disorders.
* History of severe diseases involving heart, kidney, marrow, lung or central neural system.
* Infection diseases which need antibiotics treatment before less than 1 month.
* Co-existing morbidity or social environment which may lead patients not to obey study protocol or threat patients' safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) of intrahepatic lesions | 2 years
  Assess the Disease control rate (DCR) of intrahepatic lesions by enhanced CT or MRI scan according to RECIST criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | 30 month
  From the date of first D-TACE to the date of death from any cause or to completion of trial, whichever comes first, up to 30 months.
Progression Free Survival (PFS) | 30 months
  From the date of first D-TACE to the date of documented disease progression, including progression of intrahepatic lesions and progression of extrahepatic lesions, or to completion of trial, whichever comes first, up to 30 months.
Quality of life (QOL) | 30 months
  Assessed according to EORTC QLQ-C30(V3.0)
Side effects and adverse events | 30 months
  To determine the safety and tolerability of DEBOXA for NEN liver metastases

CONTACTS AND LOCATIONS:
Overall Officials: Liangrong Shi, M.D., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China